CLINICAL TRIAL: NCT00772720
Title: Study on the Effects of Raltegravir (Isentress®) on Lipid and Carbohydrate Metabolism and Mitochondrial Function in Healthy Volunteers
Brief Title: Effects of Raltegravir (Isentress®) on Lipid and Carbohydrate Metabolism and Mitochondrial Function in Healthy Volunteers
Acronym: RALMET-VOLHCB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Jose M Gatell, Hospital Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RALMET-VOLHCB; EUDRACT #: 2008- 003288-37
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: raltegravir — raltegravir 400 mg BID for 7 days
  Other Names: Isentress
Drug: Placebo — Placebo BID for 7 days

SUMMARY:
Raltegravir is the first of a new antiretroviral class. A better profile of metabolic toxicity is expected. In order to better define its effects, without interference with other drugs, a study on healthy volunteers is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male.
2. age between 18 and 45.
3. BMI between 19 and 25 kg/m2
4. Normal physical exam.
5. Blood analysis without relevant findings.
6. Negative serology for hepatitis B, Hepatitis C and HIV.
7. Negative urine test for abuse drugs.

Exclusion Criteria:

1. Severe psychiatric disease.
2. Dyslipemia.
3. Alcohol intake above 30 g per day.
4. Smokers
5. Xanthine intake above 5 coffee cup -equivalents per day
6. Use of any drugs in the last month
7. Participation in other trials in the last 3 months
8. Diseases capable to modify drug ADME
9. Drug allergy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Blood levels of total cholesterol | 7 days

SECONDARY OUTCOMES:
Changes in HDL, LDL and triglycerides | 7 days
Oral glucose tolerance test | 7 days
Mitochondrial DNA levels | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain